CLINICAL TRIAL: NCT05438394
Title: Clinical Study of Safety and Tolerability of Melphalan Hydrochloride for Injection in the Treatment of Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Clinical Study of Safety and Tolerability of Melphalan Hydrochloride for R/R MM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, JinLu, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021PHD013-001
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Injections

STUDY DESIGN:
Intervention Model Description: Four dose groups. Using the "3 + 3" dose escalation principle, 3-6 subjects per dose group, according to the dose limiting toxicity (DLT) observed in the first cycle of chemotherapy for each subject. After completing the 21-day assessment of the first cycle of chemotherapy, if there was no DLT, the study started for the next dose group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- melphalan hydrochloride for injection (Experimental): Drug Name: melphalan hydrochloride The dosage of different dosage groups were: 9 mg/m2; 18 mg/m2; 27 mg/m2; 40 mg/m2 Administration frequency: once for each subject
  Interventions: Drug: melphalan hydrochloride for injection

INTERVENTIONS:
Drug: melphalan hydrochloride for injection — Intravenous (iv) infusion for 20 minutes on Day 1 of a 21-day chemotherapy cycle

SUMMARY:
This study is an investigator-initiated clinical study to evaluate the safety and tolerability of melphalan hydrochloride for injection in patients with relapsed or relapsed refractory multiple myeloma. Using the "3 + 3" dose escalation principle, 3-6 subjects per dose were enrolled, depending on the dose limiting toxicity (DLT) observed in the first cycle of chemotherapy for each subject. After completing the 21-day assessment of the first cycle of chemotherapy, if there was no DLT, the study started for the next dose group.

DETAILED DESCRIPTION:
The escalation method was as follows: 1 subject in each dose group was evaluated for safety by the investigator, and another 2 subjects were evaluated with the permission of the investigator: if none of them experienced DLT, they were escalated to the next dose group.If 1 subject experiences DLT, another 3 subjects will be enrolled in the same dose group.If DLT is not observed in 3 newly added subjects, the study of the next dose group can be started.Dose escalation was terminated if 2 or more DLTs were observed in 3 subjects enrolled in each dose group, or 1 or more DLTs were observed in 3 additional subjects per group.This dose was judged as "intolerable dose", and dose escalation was stopped at the same time. The previous dose group was used as MTD. If only 3 patients were enrolled in the previous dose group, 3 more patients were required (the continued dose escalation should be less than"intolerable dose"). DLT was continued to be observed to determine MTD. Dose escalation for the same subject was not permitted.If a subject dropped out during the DLT observation period due to non-DLT reasons or did not complete DLT observation according to the protocol, continued enrollment of subjects is required to meet the requirement of 3 or 6 subjects per dose. The administration method is as follows: Melphalan Hydrochloride for Injection 9 mg/m2, 18 mg/m2, 27 mg/m2 and 40 mg/m2 (if there is no DLT in this dose group when the dose is up to 40 mg/m2).The primary objective of this phase is to determine the optimal dose of melphalan hydrochloride for injection, up to 40 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female;
2. Relapsed or refractory multiple myeloma according to IMWG. There is no requirement for the number of previous treatment lines in this study
3. With any one of the following measurable indicators: serum protein electrophoresis (SPEP) ≥ 1 g/dL (10 g/L), if IgA, IgD, IgE or IgM multiple myeloma subjects, ≥ 0.5 g/dL (≥ 5 g/L); urine M protein ≥ 200 mg/24h; serum free light chain (FLC) ≥ 10 mg/dL and abnormal serum free light chain kappa/lambda ratio;
4. Life expectancy ≥ 6 months;
5. ECOG score ≤ 2;
6. ECG QT interval ≤ 470 ms;
7. Neutrophil ≥ 1.0*10^9/L, platelet ≥ 75*10^9/L (or 50 *10^9/L if plasma cell infiltration in bone marrow more than 50%);
8. Tbil ≤1.5 ULN，AST and ALT≤3.0 ULN （Gilbert syndrome except);
9. eGFR ≥ 45 ml/min or creatinine ≤ 2mg/dl
10. Understand the contents of this study and have signed the informed consent form.

Exclusion Criteria:

1. primary amyloidosis, MGUS, or smoldering multiple myeloma or plasma cell leukemia (according to the World Health Organization criteria: peripheral blood ≥ 5%) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin) ;
2. primary refractory disease (i.e., no at least MR response to any prior therapy);
3. combined clinically significant comorbidities (investigator judged);
4. the presence of active infection;
5. history of other malignant tumors (except multiple myeloma) within 3 years before signing the informed consent;
6. Pregnant or lactating women;
7. radiotherapy or other anti-myeloma treatment within 14 days before signing the informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | one month
  Hematological toxicity: Grade 4 thrombocytopenia OR Grade 4 neutropenia more than 7 days; Any non - hematological toxicity of grade 3 or above, except: 1) Grade 3 nausea / vomiting or diarrhea with duration less than 72 hours; 2) Grade 3 fatigue with duration less than one week; Grade 3 fever; Grade 4 infusion reaction;

SECONDARY OUTCOMES:
The overall response rate | one month
  Hematological response CR + VGPR + PR +MR
TTP | 12 months
  Time to progression
Progression-Free Survival (PFS) | 12 months
  PFS is defined as the time from drug administration to progression or death, whichever occurs first
Overall Survival (OS) | 12 months
  OS is defined as the time from drug administration to death.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No